CLINICAL TRIAL: NCT05950035
Title: An Efficient Treatment for Posttraumatic Injury for Firefighters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: University of Arizona (Other); Oregon State University (Other); Boston University (Other); The University of Texas Health Science Center at San Antonio (Other); National Development and Research Institutes, Inc. (Other)
Responsible Party: Principal Investigator, Carmen McLean, Clinical Psychologist, Palo Alto Veterans Institute for Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MCA0006AGG
Record Dates: First submitted 2023-06-05; First posted 2023-07-18 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Posttraumatic Stress Disorder; Insomnia; Nightmare
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy; Waiting Lists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Intervention (Experimental): Will begin treatment within 2 weeks of randomization.
  Interventions: Behavioral: Written Exposure Therapy (WET); Behavioral: Cognitive Behavioral Therapy for Insomnia (CBTi); Behavioral: Cognitive Behavioral Therapy for Nightmares (CBTn)
- Delayed Intervention (Active Comparator): Will be scheduled to begin treatment within 4-6 weeks of randomization.
  Interventions: Behavioral: Waitlist

INTERVENTIONS:
Behavioral: Written Exposure Therapy (WET) — WET is a trauma-focused intervention in which individuals write about their worst traumatic experience following scripted instruction from the therapist.
  Arms: Immediate Intervention
Behavioral: Cognitive Behavioral Therapy for Insomnia (CBTi) — CBTi focuses on stimulus control, eliminating maladaptive coping habits, reducing arousal, and challenging maladaptive thoughts about sleep in an effort to reduce time to fall asleep and time awake during the night.
  Arms: Immediate Intervention
Behavioral: Cognitive Behavioral Therapy for Nightmares (CBTn) — CBTn involves writing about a distressing or frequent nightmare, rewriting the narrative of the nightmare to target trauma-related themes, and reading the rescripted nightmare narrative.
  Arms: Immediate Intervention
Behavioral: Waitlist — Waitlist for delayed intervention.
  Arms: Delayed Intervention

SUMMARY:
The goal of this two-arm pilot randomized controlled trial is to test a behavioral intervention that integrates three evidence-based cognitive behavioral interventions (written exposure therapy; WET, cognitive behavioral therapy for insomnia; CBT-I, and cognitive behavioral therapy for nightmares; CBT-N) among firefighters. The main questions it aims to answer are:

* Is the behavioral intervention feasible, acceptable, and effective in reducing symptoms of posttraumatic stress, insomnia, and nightmares?
* What is the efficacy of efficient treatment vs. delayed treatment (2-4 week waitlist) in reducing symptoms of posttraumatic stress, insomnia, and nightmares?

We will beta test the intervention in 1-2 groups of 3-5 firefighters. Then we will randomize 50 participants to immediate or delayed (2-4 week waitlist) treatment. Consented participants will:

* Complete self-report and interview measures assessing posttraumatic stress disorder, insomnia (PTSD), and nightmares
* Attend an individual treatment orientation session
* Attend a 4-day (~3 hours per day over 4 consecutive days) group treatment that integrates WET, CBT-I, and CBT-N
* Attend an individual booster session held approximately one week later
* Complete self-report measures before, during, and after treatment, and at a 3-month follow up assessment and a clinical interview before and after treatment to assess program efficacy.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Firefighter
* Able to speak and read English
* Clinically significant posttraumatic stress symptoms: CAPS-5 total score ≥ 25; ≥ 1 intrusion symptom; ≥ 1 avoidance symptom
* Clinically significant symptoms of insomnia: SCISD insomnia criteria are met; ISI ≥ 15
* Clinically significant symptoms of nightmare disorder: SCISD nightmare disorder criteria are met, nightmares ≥ 1 monthly.

Exclusion Criteria:

* Current suicide or homicide risk meriting crisis intervention
* Inability to speak and read English
* Inability to comprehend the baseline screening questionnaires
* Unwilling to remain abstinent from alcohol during treatment
* Serious mental health diagnosis such as bipolar disorder or psychosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS-5) | Change from baseline to post treatment (~4 weeks post baseline)
  The CAPS-5 is a structured clinical interview that assesses the presence and severity of PTSD symptoms.
Structured Clinical Interview for DSM-5 Sleep Disorders- Revised (SCISD-R) | Change from baseline to post treatment (~4 weeks post baseline)
  The SCISD-R is a semi-structured interview designed to obtain a sleep history and screen for certain sleep disorders and diagnose others, including insomnia, hypersomnia, circadian rhythm sleep-wake disorders, sleep-disordered breathing, and parasomnias.
Insomnia Severity Index (ISI) | Change from baseline through 3 months post treatment
  The ISI assesses perceived severity of insomnia.
Nightmare Disorders Index | Change from baseline through 3 months post treatment
  The NDI is a self-report assessment of nightmare disorder.
Posttraumatic Stress Disorder Checklist (PCL-5) | Change from baseline through 3 months post treatment
  Self-report measure update of the PCL designed to assess PTSD symptoms as defined by the DSM-5.

SECONDARY OUTCOMES:
Trauma-Related Nightmare Survey (TRNS) | Change from baseline through 3 months post treatment
  The TRNS assesses nightmare frequency, disturbance, and characteristics.
Self-Assessment of Sleep (SASS) | Change from baseline through 3 months post treatment
  The SASS is a brief assessment of self-reported sleep quantity and sleep quality.
Sleep Diary and Nightmare Log | Change from baseline through post treatment (~4 weeks post baseline)
  The Sleep Diary and Nightmare Log assess daily subjective sleep patterns and to inform treatment recommendations.
Patient Health Questionnaire-9 (PHQ-9) | Change from baseline through 3 months post treatment
  The PHQ-9 the severity of affective and somatic symptoms related to depression; items correspond to the diagnostic criteria for major depression disorder.
Depressive Symptoms Index-Suicidality Subscale (DSI-SS) | Change from baseline through 3 months post treatment
  The DSI-SS is a self-report measure of suicidal ideation, plans, perceived control over ideation, and impulses for suicide.
Net Prompter Score | Post treatment (~4 weeks post baseline)
  The Net Prompter Score is a single item measures of treatment acceptability that asks respondents to rate the likelihood that they would recommend the efficient treatment to a friend or colleague on a scale from 0-10.

CONTACTS AND LOCATIONS:
Locations (1):
- NDRI_USA, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McLean CP, Janke S, Pruiksma KE, Taylor DJ, Sloan DM, Dietch JR, Fredman SJ, Sutherland C, Hollerbach B, Thompson SM, Tse D, Nagy S, Malek N, Haddock CK. A pilot feasibility randomized clinical trial of a culturally adapted accelerated group treatment for posttraumatic stress, insomnia, and nightmares in firefighters. Psychol Trauma. 2026 Jan 19. doi: 10.1037/tra0002090. Online ahead of print. PMID 41556892